CLINICAL TRIAL: NCT04934449
Title: The Effect of Occlusal Splint Type on Sleep Quality and Occlusal Force in Patients With Sleep Bruxism
Brief Title: Occlusal Splints in the Treatment of Sleep Bruxism
Acronym: bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1299
Record Dates: First submitted 2021-06-16; First posted 2021-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Sleep Bruxism, Adult; Splints; Sleep
Keywords: sleep quality; occlusal splint; bruxism
MeSH Terms: conditions — Sleep Bruxism; Sleep Initiation and Maintenance Disorders; Bruxism | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Blinding the participants and investigator to the splint types employed in patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hard splint group- 2 mm thicknesss (Experimental): This group of patients was allocated to use 2 mm-thickness, hard occlusal splints for 2 months during sleep
  Interventions: Device: Occlusal splint
- Hard splint group- 3 mm thicknesss (Experimental): This group of patients was allocated to use 3 mm-thickness, hard occlusal splints for 2 months during sleep
  Interventions: Device: Occlusal splint
- Soft splint group- 2 mm thicknesss (Experimental): This group of patients was allocated to use 2 mm-thickness, soft occlusal splints for 2 months during sleep
  Interventions: Device: Occlusal splint
- Soft splint group- 3 mm thicknesss (Experimental): This group of patients was allocated to use 3 mm-thickness, soft occlusal splints for 2 months during sleep
  Interventions: Device: Occlusal splint

INTERVENTIONS:
Device: Occlusal splint — Using occlusal splints during sleep for 2 months

SUMMARY:
Occlusal splints are employed in the treatment of sleep bruxism. These appliances decrease sleep-related actions and damages bruxism, like grinding, tooth-wear, headache, and temporomandibular joint disorders. Occlusal splints are produced both in hard and soft forms according to the used material.

In this study, it was aimed to evaluate the effect of occlusal splint type on the sleep quality and occlusal force parameters of patients with sleep bruxism.

DETAILED DESCRIPTION:
Various splint designs have been used for the treatment of sleep bruxism that is made up of different materials: Hard and soft splints. Although, these splints have slightly different appearances and properties, in fact, scientific evidence supports both the use of hard and soft occlusal splints. Hard splints are more preferred when compared to soft ones, thus, oft appliances have been less documented in the scientific literature. However, some studies suggested the use of soft-resin splints that are easily fabricated and may be inserted at an initial appointment, dental clinicians may desire the use of soft appliances. One of the advantages of these appliances is they are easy to tolerable to the patient and comfortable. Additionally, these splints fit tightly and provide a flat plane during sleep.

Considering these advantages, the present study was designed to examine the effect of the use of different types of occlusal splints on the sleep quality and occlusal force of patients with sleep bruxism. For this purpose, the effect of two splints basically fabricated from two different materials were evaluated and compared. The null hypothesis was that the use of both occlusal splints would not change the values of sleep quality and maximum occlusal force of the patients with sleep bruxism.

ELIGIBILITY:
Inclusion Criteria:

- Healthy participants with complete permanent dentition.

Exclusion Criteria:

* Presence of a systemic disorder that could compromise the masticatory system (e.g., neurological disorders, epilepsy, cerebral palsy, among others),
* Systemic disorder or current use of drugs that could interfere, directly or indirectly, with muscle activity,
* Inappropriate behavior and/or refusal to cooperate with dental procedures and data collection,
* Tooth loss (except for third molars),
* Soft tissue abnormalities,
* Toothache report,
* Active periodontitis (presence of periodontal pockets involvement of the supporting tissues),
* Caries lesions,
* Use of orthodontic appliances,
* Use of dental prosthesis (fixed or removable partial).
* Subjects with moderate to severe malocclusions, diagnosed by using the Orthodontic Treatment Need Index (IOTN) (scores 5 or 6 - severe and extreme need for orthodontic treatment)
* Alcohol or drug abuse,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 2 months
  Evaluating sleep quality with Pittsburgh sleep quality index
occlusal force | 2 months
  Measuring maximum occlusal force by using digital gnatodynanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university,Faculty of Dentistry, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosar JV, Barbosa TS, Dias IOV, Kobayashi FY, Costa YM, Gaviao MBD, Bonjardim LR, Castelo PM. Effect of interocclusal appliance on bite force, sleep quality, salivary cortisol levels and signs and symptoms of temporomandibular dysfunction in adults with sleep bruxism. Arch Oral Biol. 2017 Oct;82:62-70. doi: 10.1016/j.archoralbio.2017.05.018. Epub 2017 May 27. PMID 28601734